CLINICAL TRIAL: NCT01073293
Title: A Phase III Open-Label Clinical Trial to Study the Immunogenicity and Tolerability of V503, a Multivalent Human Papillomavirus (HPV) L1 Virus-Like Particle (VLP) Vaccine, Given Concomitantly With REPEVAX™ in Preadolescents and Adolescents (11 to 15 Year Olds)
Brief Title: A Study of V503 Vaccine Given Concomitantly With REPEVAX™ in 11 to 15 Year Olds (V503-007)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V503-007; 2010_512 (Other Grant/Funding Number: Merck Registration Number)
Record Dates: First submitted 2010-02-19; First posted 2010-02-23 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-10

CONDITIONS: Papillomavirus Infections
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concomitant Vaccination (Experimental): V503 given as a 0.5 mL intramuscular injection in the deltoid muscle of the non-dominant arm on Day 1, Month 2, and Month 6, and Repevax™ given as a 0.5 mL intramuscular injection in the deltoid muscle of the dominant arm on Day 1
  Interventions: Biological: V503 Vaccine; Biological: REPEVAX™ (Concomitant)
- Non-concomitant Vaccination (Experimental): V503 given as a 0.5 mL intramuscular injection in the deltoid muscle of the non-dominant arm on Day 1, Month 2, and Month 6, and Repevax™ given as a 0.5 mL intramuscular injection in the deltoid muscle of the dominant arm at Month 1
  Interventions: Biological: V503 Vaccine; Biological: REPEVAX™ (Non-concomitant)

INTERVENTIONS:
Biological: V503 Vaccine — V503 (Multivalent HPV L1 VLP vaccine) given as a 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6
Biological: REPEVAX™ (Concomitant) — REPEVAX™ given as a single 0.5 mL intramuscular injection at Day 1
  Arms: Concomitant Vaccination
Biological: REPEVAX™ (Non-concomitant) — REPEVAX™ given as a single 0.5 mL intramuscular injection at Month 1
  Arms: Non-concomitant Vaccination

SUMMARY:
This study will evaluate whether co-administration of the first dose of V503 and REPEVAX™ is well tolerated and causes a non-inferior immune response when compared to administration of REPEVAX™ one month following the first dose of V503.

ELIGIBILITY:
Inclusion criteria:

* Participant is in good health
* Participant's parent/legal guardian can read, understand, and complete the vaccination report card
* Participant is not sexually active and does not plan on becoming sexually active during the study
* Participant has received a documented full primary immunization series against diphtheria, tetanus, pertussis, and poliovirus (inactivated and/or oral poliovirus), but not in the last 5 years. There must be a 5-year interval from a prior vaccination containing any one of these vaccine antigens.

Exclusion Criteria:

* Participant has a known allergy to any vaccine component of V503 or REPEVAX™
* Participant has had a severe reaction affecting the brain (e.g., evolving encephalopathy) within 7 days after a previous dose of a pertussis-containing vaccine
* Participant has had a progressive severe illness affecting the brain after a previous dose of tetanus, diphtheria, poliovirus or a component pertussis combination (acellular and whole cell) vaccine
* Participant ever had Guillain-Barré syndrome or brachial neuritis following a previous dose of a tetanus-containing vaccine
* Participant has a condition that is a contraindication to vaccination as indicated in the most up to date package inserts of REPEVAX™
* Participant has a history of severe allergic reaction that required medical intervention
* Participant has hemophilia, thrombocytopenia, is receiving anticoagulation therapy and/or has any coagulation disorder that would contraindicate intramuscular injections
* Participant is concurrently enrolled in clinical studies of investigational agents
* Female participant is pregnant
* Participant has donated blood within 1 week prior to first study vaccination, or intends to donate during the study
* Participant is immunocompromised, immunodeficient, or has an autoimmune condition
* Participant has had a splenectomy
* Participant has received immunosuppressive therapies in the prior year
* Participant has received immune globulin product or blood-derived product in the last 3 months
* Participant has received inactivated vaccine(s) within 14 days or live vaccine(s) within 21 days of first study vaccination
* Participant has received a marketed HPV vaccine or has participated in an HPV vaccine trial
* Participant has received a tetanus, diphtheria, pertussis, or poliovirus (inactivated and/or oral poliovirus) vaccination within the last 5 years
* Participant has a fever ≥100°F within 24 hours of vaccination
* Participant has any history or current condition, therapy, lab abnormality, or other circumstance such that it is not in the best interest of the participant to participate
* Participant and parent/legal guardian are unable to give assent/consent
* Participant is unlikely to adhere to the study procedures or is planning to relocate during the study
* Participant has recent history of illicit drug or alcohol abuse
* Participant has a history of HPV

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1054 (Actual)
Dates: Start 2010-04-22 (Actual); Primary Completion 2011-06-16 (Actual); Study Completion 2011-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Kosalaraksa P, Mehlsen J, Vesikari T, Forsten A, Helm K, Van Damme P, Joura EA, Ciprero K, Maansson R, Luxembourg A, Sobanjo-ter Meulen A. An open-label, randomized study of a 9-valent human papillomavirus vaccine given concomitantly with diphtheria, tetanus, pertussis and poliomyelitis vaccines to healthy adolescents 11-15 years of age. Pediatr Infect Dis J. 2015 Jun;34(6):627-34. doi: 10.1097/INF.0000000000000694. PMID 25831420
- [Result] Moreira ED Jr, Block SL, Ferris D, Giuliano AR, Iversen OE, Joura EA, Kosalaraksa P, Schilling A, Van Damme P, Bornstein J, Bosch FX, Pils S, Cuzick J, Garland SM, Huh W, Kjaer SK, Qi H, Hyatt D, Martin J, Moeller E, Ritter M, Baudin M, Luxembourg A. Safety Profile of the 9-Valent HPV Vaccine: A Combined Analysis of 7 Phase III Clinical Trials. Pediatrics. 2016 Aug;138(2):e20154387. doi: 10.1542/peds.2015-4387. Epub 2016 Jul 15. PMID 27422279
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=V503-007&kw=V503-007&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Started | 526 | 528
Completed | 521 | 517
Not Completed | 5 | 11
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 5 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination | Total
Number analyzed (Participants) | 526 | 528 | 1054
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.4 (1.2) | 12.4 (1.2) | 12.4 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 264 | 264 | 528
  Male | 262 | 264 | 526

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of the Antibody Response to Each of the Human Papillomavirus (HPV) Types Contained in V503
Description: Serum antibody titers for HPV types 6, 11, 16, 18, 31, 33, 45, 52, and 58 were measured using a competitive Luminex immunoassay. Titers are reported in milli Merck Units/mL.
Time Frame: 4 weeks following Month 6 vaccination
Population: The per-protocol population included participants who received all study vaccinations, were seronegative to HPV on Day 1, and had serum samples available for evaluation of the endpoint
Measure: Geometric Mean (Full Range); unit: milli Merck Units/mL
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Number analyzed (Participants) | 525 | 528
milli Merck Units/mL
  Anti-HPV 6: n=477, 461 | 1637.9 [8.0 to 24405.0] | 1725.0 [173.0 to 12040.0]
  Anti-HPV 11: n=479, 462 | 1170.3 [84.0 to 13438.0] | 1212.6 [153.0 to 9816.0]
  Anti-HPV 16: n=489, 479 | 6529.4 [689.0 to 76781.0] | 6940.6 [841.0 to 49390.0]
  Anti-HPV18: n=486, 475 | 1854.1 [81.0 to 38887.0] | 1954.8 [49.0 to 15582.0]
  Anti-HPV 31: n=485, 473 | 1646.2 [88.0 to 22848.0] | 1750.6 [118.0 to 32822.0]
  Anti-HPV 33: n=487, 478 | 823.8 [54.0 to 6563.0] | 915.5 [110.0 to 7058.0]
  Anti-HPV 45: n=489, 478 | 658.2 [28.0 to 14131.0] | 675.6 [29.0 to 8725.0]
  Anti-HPV 52: n=490, 479 | 965.4 [45.0 to 11730.0] | 1015.3 [79.0 to 14392.0]
  Anti-HPV 58: n=484, 469 | 1188.8 [102.0 to 13681.0] | 1334.8 [106.0 to 14752.0]
Statistical Analysis 1: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-HPV 6; Test type: Non-Inferiority or Equivalence — Noninferiority of concomitant versus non-concomitant vaccination is demonstrated if the lower limit of the 95% confidence interval for the fold difference is >0.5; p < 0.001, ANOVA; Fold difference in GMT = 0.95, 95% CI 2-sided [0.86 to 1.05]
Statistical Analysis 2: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-HPV 11; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; Fold difference in GMT = 0.97, 95% CI 2-sided [0.87 to 1.07]
Statistical Analysis 3: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-HPV 16; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; Fold difference in GMT = 0.94, 95% CI 2-sided [0.85 to 1.04]
Statistical Analysis 4: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-HPV 18; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; Fold difference in GMT = 0.95, 95% CI 2-sided [0.84 to 1.07]
Statistical Analysis 5: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-HPV 31; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; Fold difference in GMT = 0.94, 95% CI 2-sided [0.84 to 1.06]
Statistical Analysis 6: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-HPV 33; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; Fold difference in GMT = 0.90, 95% CI 2-sided [0.81 to 1.00]
Statistical Analysis 7: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-HPV 45; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; Fold difference in GMT = 0.97, 95% CI 2-sided [0.86 to 1.11]
Statistical Analysis 8: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-HPV 52; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; Fold difference in GMT = 0.95, 95% CI 2-sided [0.85 to 1.06]
Statistical Analysis 9: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-HPV 58; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; Fold difference in GMT = 0.89, 95% CI 2-sided [0.80 to 0.99]

2. Primary Outcome: Percentage of Participants With a V503 Injection-site Adverse Experience
Description: An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the vaccine. Any worsening of a preexisting condition which is temporally associated with the use of the vaccine is also an AE. Only injection-site AEs in the arm that received V503 vaccination were reported for this endpoint.
Time Frame: Day 1 through Day 5 following Day 1 vaccination
Population: The population analyzed included all vaccinated participants with follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Number analyzed (Participants) | 524 | 527
Percentage of participants | 63.4 | 62.8

3. Primary Outcome: Percentage of Participants With a Repevax™ Injection-site Adverse Experience
Description: For the Concomitant Vaccination group, injection-site AEs are reported following Day 1 vaccination; for the Non-concomitant Vaccination group, injection-site AEs are reported following Month 1 vaccination. An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the vaccine. Any worsening of a preexisting condition which is temporally associated with the use of the vaccine is also an AE. Only injection-site AEs in the arm that received Repevax™ vaccination were reported for this endpoint.
Time Frame: Day 1 through Day 5 following Day 1 (Concomitant) or Month 1 (Non-concomitant) vaccination
Population: The population analyzed included all vaccinated participants with follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Number analyzed (Participants) | 525 | 520
Percentage of participants | 88.0 | 84.6

4. Primary Outcome: Percentage of Participants With Maximum Temperature >=37.8 °C (>=100.0 °F) (Oral or Oral Equivalent)
Description: For the Concomitant Vaccination group, temperatures were collected after the Day 1 vaccination and the Month 1 visit; for the Non-concomitant Vaccination group, temperatures were collected after the Day 1 vaccination and the Month 1 vaccination.
Time Frame: Up to 5 days following the Day 1 and Month 1 vaccination / visit
Population: The population analyzed included all vaccinated participants with follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Number analyzed (Participants) | 524 | 525
Percentage of participants | 8.8 | 8.4

5. Primary Outcome: Percentage of Participants With a Systemic Adverse Experience
Description: For the Concomitant Vaccination group, systemic AEs were collected after the Day 1 vaccination and the Month 1 visit; for the Non-concomitant Vaccination group, systemic AEs were collected after the Day 1 vaccination and the Month 1 vaccination. An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body that is temporally associated with the use of the study vaccine, whether or not considered related to the use of the vaccine. Any worsening of a preexisting condition which is temporally associated with the use of the vaccine is also an adverse experience. A systemic AE was an AE that was not associated with the injection site.
Time Frame: Up to 15 days following the Day 1 and Month 1 vaccination / visit
Population: The population analyzed included all vaccinated participants with follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Number analyzed (Participants) | 525 | 527
Percentage of participants | 48.6 | 48.6

6. Primary Outcome: Percentage of Participants Who Achieve Acceptable Titers of Anti-Diphtheria and Anti-Tetanus Antibody
Description: For the Concomitant Vaccination group, serum samples were collected 4 weeks after the Day 1 vaccination; for the Non-concomitant Vaccination group, serum samples were collected 4 weeks after the Month 1 vaccination. Titers of neutralizing antibody to diphtheria toxin were measured using a cell-based Diphtheria Micrometabolic Inhibition assay. Serum titers of neutralizing antibody to tetanus toxin were measured using an enzyme immunoassay. The lower limits of quantitation of the assays was 0.01 International Units (IU)/mL and 0.04 IU/mL, respectively. Acceptable titers refer to the World Health Organization-defined protective titer of >=0.1 IU/mL.
Time Frame: 4 weeks following Day 1 (Concomitant) or Month 1 (Non-concomitant) vaccination
Population: The per-protocol population included participants who received vaccination and had serum samples available for evaluation of the endpoint
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Number analyzed (Participants) | 525 | 528
Percentage of participants
  Anti-diphtheria titer >=0.1 IU/mL: n=505, 474 | 99.8 [98.9 to 100] | 99.6 [98.5 to 99.9]
  Anti-tetanus titer >=0.1 IU/mL: n=504, 472 | 99.6 [98.6 to 100] | 99.6 [98.5 to 99.9]
Statistical Analysis 1: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-diphtheria titer >=0.1 IU/mL; Test type: Non-Inferiority or Equivalence — Noninferiority of concomitant versus non-concomitant vaccination is demonstrated if the lower limit of the 95% confidence interval for the percentage difference is greater than -10; p < 0.001, Miettinen and Nurminen; Difference in percentage = 0.2, 95% CI 2-sided [-0.7 to 1.4]
Statistical Analysis 2: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-tetanus titer >=0.1 IU/mL; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in percentage = 0.0, 95% CI 2-sided [-1.1 to 1.2]

7. Primary Outcome: Geometric Mean Titers of Pertussis Antibody Responses
Description: For the Concomitant Vaccination group, serum samples were collected 4 weeks after the Day 1 vaccination; for the Non-concomitant Vaccination group, serum samples were collected 4 weeks after the Month 1 vaccination. Titers of anti-pertussis toxin (PT), anti-filamentous hemagglutinin (FHA), anti-pertactin (PRN), and anti-fimbriae 2/3 (FM 2/3) antibodies were measured using enzyme-linked immunosorbent assays. Titers are expressed as enzyme-linked immunoassay units/mL (ELU/mL).
Time Frame: 4 weeks following Day 1 (Concomitant) or Month 1 (Non-concomitant) vaccination
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ELU/mL
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Number analyzed (Participants) | 525 | 528
ELU/mL
  Anti-PT: n=505, 473 | 41.5 [38.4 to 44.9] | 43.8 [40.4 to 47.5]
  Anti-FHA: n=505, 474 | 188.1 [176.2 to 200.8] | 190.6 [178.1 to 203.9]
  Anti-PRN: n=505, 474 | 372.9 [334.8 to 415.2] | 398.2 [356.3 to 445.0]
  Anti-FIM 2/3: n=505, 474 | 378.2 [324.4 to 440.9] | 423.6 [361.5 to 496.2]
Statistical Analysis 1: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-PT; Test type: Non-Inferiority or Equivalence — Noninferiority of concomitant versus non-concomitant vaccination is demonstrated if the lower limit of the 95% confidence interval for the fold difference is >0.67; p < 0.001, ANOVA; Fold difference in GMT = 0.95, 95% CI 2-sided [0.85 to 1.06]
Statistical Analysis 2: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-FHA; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 7, analysis 1]; p < 0.001, ANOVA; Fold difference in GMT = 0.99, 95% CI 2-sided [0.90 to 1.08]
Statistical Analysis 3: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-PRN; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 7, analysis 1]; p < 0.001, ANOVA; Difference in GMT = 0.94, 95% CI 2-sided [0.80 to 1.09]
Statistical Analysis 4: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-FIM 2/3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 7, analysis 1]; p = 0.005, ANOVA; Difference in GMT = 0.89, 95% CI 2-sided [0.72 to 1.11]

8. Primary Outcome: Percentage of Participants Who Achieve Acceptable Titers of Anti-Poliovirus Antibody
Description: For the Concomitant Vaccination group, serum samples were collected 4 weeks after the Day 1 vaccination; for the Non-concomitant Vaccination group, serum samples were collected 4 weeks after the Month 1 vaccination. Titers of neutralizing antibody to poliovirus type 1, 2, and 3 were measured using a microneutralization assay. Serial dilutions of sera were incubated with type-specific standard poliovirus and sensitive cells. Neutralization of the virus was measured by cell staining. Acceptable titers were defined as neutralization at >=1:8 dilution of serum.
Time Frame: 4 weeks following Day 1 (Concomitant) or Month 1 (Non-concomitant) vaccination
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Number analyzed (Participants) | 525 | 528
Percentage of participants
  Poliovirus type 1: n=505, 474 | 99.6 [98.4 to 100] | 99.8 [98.7 to 100]
  Poliovirus type 2: n=505, 474 | 99.6 [98.4 to 100] | 99.8 [98.7 to 100]
  Poliovirus type 3: n=505, 474 | 100 [99.1 to 100] | 100 [99.1 to 100]
Statistical Analysis 1: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Poliovirus type 1; Test type: Non-Inferiority or Equivalence — Noninferiority of concomitant versus non-concomitant vaccination is demonstrated if the difference is statistically less than 10 percentage points; p < 0.001, Miettinen and Nurminen; Difference in percentage = -0.2, 95% CI 2-sided [-1.2 to 0.8]
Statistical Analysis 2: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Poliovirus type 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 8, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in percentage = -0.2, 95% CI 2-sided [-1.2 to 0.8]
Statistical Analysis 3: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Poliovirus type 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 8, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in percentage = 0.0, 95% CI 2-sided [-0.8 to 0.8]

9. Secondary Outcome: Percentage of Participants Who Seroconvert for Each of the HPV Types
Description: Blood was drawn at Month 7 and assayed to determine whether or not a participant had achieved seroconversion for the HPV types. The lower limit of the titer (milli Merck U/mL) considered seropositive was as follows: HPV Type 6: >=30, HPV Type 11: >=16; HPV Type 16: >=20, HPV Type 18: >=24, HPV Type 31: >=10, HPV Type 33: >=8, HPV Type 45: >=8, HPV Type 52: >=8, and HPV Type 58: >=8.
Time Frame: Month 7
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Number analyzed (Participants) | 525 | 528
Percentage of participants
  Anti-HPV 6: n=477, 461 | 99.8 | 100.0
  Anti-HPV 11: n=479, 462 | 100.0 | 100.0
  Anti-HPV 16: n=489, 479 | 100.0 | 100.0
  Anti-HPV 18: n=486, 475 | 100.0 | 100.0
  Anti-HPV 31: n=485, 473 | 100.0 | 100.0
  Anti-HPV 33: n=487, 478 | 100.0 | 100.0
  Anti-HPV 45: n=489, 478 | 100.0 | 100.0
  Anti-HPV 52: n=490, 479 | 100.0 | 100.0
  Anti-HPV 58: n=484, 469 | 100.0 | 100.0

ADVERSE EVENTS:
Time Frame: Serious adverse events: up to Month 7; Other adverse events: Day 1 through Day 5 following any vaccination for injection-site AEs and Day 1 through Day 15 following any vaccination for non-injection-site AEs
Description: Adverse events were collected for all participants who received at least one dose of V503 and Repevax™
Groups:
- Concomitant Vaccination: V503 given as a 0.5 mL intramuscular injection in the deltoid muscle of the non-dominant arm on Day 1, Month 2, and Month 6, and Repevax™ given as a 0.5 mL intramuscular injection in the deltoid muscle of the dominant arm at Day 1
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Serious Adverse Events (participants affected / at risk) | 9/525 | 7/527
Other Adverse Events (participants affected / at risk) | 509/525 | 505/527
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concomitant Vaccination (N=525) | Non-concomitant Vaccination (N=527)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 2 (2)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Eating disorder (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concomitant Vaccination (N=525) | Non-concomitant Vaccination (N=527)
Abdominal pain upper (Gastrointestinal disorders) | 19 (22) | 28 (28)
Nausea (Gastrointestinal disorders) | 39 (42) | 36 (46)
Injection-site erythema (General disorders) | 228 (351) | 185 (290)
Injection-site pain (General disorders) | 501 (1500) | 493 (1463)
Injection-site pruritus (General disorders) | 28 (31) | 27 (36)
Injection-site swelling (General disorders) | 295 (528) | 230 (403)
Pyrexia (General disorders) | 88 (105) | 71 (86)
Nasopharyngitis (Infections and infestations) | 18 (18) | 32 (39)
Upper respiratory tract infection (Infections and infestations) | 23 (24) | 27 (31)
Headache (Nervous system disorders) | 167 (265) | 140 (200)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 (25) | 30 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.